CLINICAL TRIAL: NCT04731675
Title: An Adaptive, Multicenter, Open-Label Study to Evaluate the Safety, Tolerability, Efficacy, and Pharmacokinetics of Intra-articular AMB-05X Injections in Subjects With Tenosynovial Giant Cell Tumor of the Knee
Brief Title: An Open-Label Study of Intra-articular AMB-05X Injections in Subjects With Tenosynovial Giant Cell Tumor of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AmMax Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMB-051-01
Record Dates: First submitted 2021-01-19; First posted 2021-02-01 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Tenosynovial Giant Cell Tumor; Pigmented Villonodular Synovitis (PVNS)
Keywords: Tenosynovial Giant Cell Tumor (TGCT); Pigmented villonodular synovitis (PVNS); TGCT; PVNS
MeSH Terms: conditions — Giant Cell Tumor of Tendon Sheath; Synovitis, Pigmented Villonodular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMB-05X (Experimental): Subjects will receive an intra-articular injection of AMB-05X once every 2 weeks for 12 weeks (for 6 treatments total).
  Interventions: Biological: AMB-05X

INTERVENTIONS:
Biological: AMB-05X — AMB-05X is a fully human antibody antagonist (immunoglobulin G, type 2 [IgG2]) specific to the extracellular domain of human CSF1R

SUMMARY:
AMB-051-01 is a multicenter study with an adaptive design that will enroll subjects with Tenosynovial Giant Cell Tumor (TGCT) of the knee for 12 weeks of multiple-dose, open-label treatment with intra-articular AMB-05X.

DETAILED DESCRIPTION:
AMB-05X drug substance is a human monoclonal antibody against the colony-stimulating factor 1 receptor (CSF1R). Study

ELIGIBILITY:
Inclusion Criteria:

1. Subject ≥ 18 years
2. A confirmed diagnosis of tenosynovial giant cell tumor (TGCT) of the knee joint
3. Measurable disease based on RECIST v1.1
4. Stable prescription of analgesic regimen
5. Negative urine drug screen (UDS) at Screening and Baseline
6. Women of childbearing potential must have a negative pregnancy test
7. Agrees to follow contraception guidelines
8. Adequate hematologic, hepatic, and renal function, at Screening
9. Willing and able to complete self-assessment instruments throughout the study

Exclusion Criteria:

1. Prior investigational drug use within 4 weeks or 5 half-lives of Baseline
2. Previous use of therapeutics targeting CSF1 or CSF1R or oral tyrosine kinase inhibitors
3. History of extensive knee surgery
4. Active cancer (either currently or within 1 year before Baseline) that requires therapy (e.g., surgery, chemotherapy, or radiation therapy)
5. Metastatic TGCT
6. Hepatitis C virus (HCV) or hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
7. Known active tuberculosis
8. Significant concomitant arthropathy in the affected joint, serious illness, uncontrolled infection, or a medical or psychiatric history
9. Women who are breastfeeding
10. A screening Fridericia-corrected QT interval (QTcF) ≥ 450 ms (men) or ≥ 470 ms (women)
11. MRI contraindications (e.g., pacemaker, loose metallic implants)
12. History of hypersensitivity to any ingredient of the study drug
13. History of drug or alcohol abuse within 3 months before the first dose of study drug
14. Any other severe acute or chronic medical or psychiatric condition or clinically significant laboratory abnormality that may increase the risk associated with study participation/treatment or interfere with interpretation of study results and, in the Investigator's opinion, make the subject inappropriate for this study
15. Subjects who, in the Investigator's opinion, should not participate in the study for any reason, including if there is a question about their ability to comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Nguyen, MD, Study Chair — AmMax Bio, Inc.
Locations (6):
- AmMax Bio Clinical Site, Columbus, Ohio, United States
- AmMax Bio Clinical Site, Leiden, Netherlands
- AmMax Bio Clinical Site, Warsaw, Poland
- Ukraine (3):
  - AmMax Bio Clinical Site, Dnipro
  - AmMax Bio Clinical Site, Kharkiv
  - AmMax Bio Clinical Site, Kyiv

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AMB-05X High Dose; ABM-05X Low Dose: Subjects with TGCT of the knee will receive an intra-articular injection of AMB-05X once every 2 weeks for 12 weeks (for 6 treatments total).
Period: Overall Study
Arm/Group | AMB-05X High Dose | ABM-05X Low Dose
Started | 8 | 3
Completed | 6 | 3
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: Subjects with TGCT of the knee
Groups:
- AMB-05X Low Dose; AMB-05X High Dose: Subjects with TGCT of the knee received an intra-articular injection of AMB-05X once every 2 weeks for 12 weeks (for 6 treatments total).
- Total: Total of all reporting groups
Arm/Group | AMB-05X Low Dose | AMB-05X High Dose | Total
Number analyzed (Participants) | 3 | 8 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 7 | 10
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 5
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 2 | 6 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Frequency and severity of reported treatment-emergent adverse events
Time Frame: 24 weeks
Population: All enrolled pts
Measure: Count of Participants; unit: Participants
Groups:
- AMB-05X - High Dose; AMB-05X Low Dose: Subjects with TGCT of the knee received an intra-articular injection of AMB-05X once every 2 weeks for 12 weeks (for 6 treatments total).
Arm/Group | AMB-05X - High Dose | AMB-05X Low Dose
Number analyzed (Participants) | 8 | 3
Participants | 7 | 2

2. Secondary Outcome: Tumor Response Based on RECIST Version 1.1
Description: Proportion of subjects who achieve an overall tumor response (Objective Response or OR) per the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 at week 12, Objective Response is defined as complete response [CR] and partial response [PR]) per RECIST v1.1 (Eisenhauer 2009) at Week 12.
  Complete response: disappearance of all target lesions; Partial Response: >/=30% decrease in the sum of diameters of target lesions.
Time Frame: Week 12
Population: All enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | AMB-05X High Dose | ABM-05X Low Dose
Number analyzed (Participants) | 8 | 3
Participants | 3 | 1

3. Secondary Outcome: Tumor Response Based on Tumor Volume (TV)
Description: Proportion of subjects with overall response based on tumor volume: Complete response (CR): lesion is completely gone; Partial response (PR): >/=50% decrease in tumor volume relative to baseline; Progressive disease (PD): >/=30% increase in tumor volume relative to the lowest volume during the study; Stable disease (SD): does not meet any of the other classifications. Tumor response based on tumor volume score ("TVS") is defined as CR or PR.
Time Frame: Week 12
Population: All enrolled patients
Measure: Count of Participants; unit: Participants
Groups:
- AMB-05X Low Dose: Subjects with TGCT of the knee will receive an intra-articular injection of AMB-05X once every 2 weeks for 12 weeks (for 6 treatments total).
Arm/Group | AMB-05X High Dose | AMB-05X Low Dose
Number analyzed (Participants) | 8 | 3
Participants | 2 | 1

4. Secondary Outcome: Mean Change From Baseline in Range of Motion (ROM): Flexion
Description: ROM of the joint will be assessed by qualified assessors. Measurements will be recorded in degrees. At baseline, the plane of movement with the smallest (worst) relative value will be identified; only this plane will be used for evaluating change in ROM subsequently.
Time Frame: Week 12
Population: All enrolled pts
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | AMB-05X High Dose | AMB-05X Low Dose
Number analyzed (Participants) | 8 | 3
degrees | 7.1 (16.3) | 3.3 (24.7)

5. Secondary Outcome: Mean Change From Baseline in the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Score
Description: The PROMIS Physical Function Scale will be used to assess physical function. The scale incudes 10 questions, with scores that range from 1 to 5, where higher scores represent better outcomes. Five questions address the degree to which the subject's health limits certain physical activities, and subjects select a response to each question that ranges from 1 ("cannot do") to 5 ("not at all"). Five additional questions address the degree to which the subject is able to perform certain physical activities, and subjects select a response to each question that ranges from 1 ("cannot do") to 5 ("without any difficulty"). The score range for the PROMIS is 10 to 50, with higher scores indicated worse physical function.
Time Frame: Week 12
Population: PROMIS Physical Function was not assessed for 1 subject in the high dose group at week 12 due to assessment not completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AMB-05X High Dose | AMB-05X Low Dose
Number analyzed (Participants) | 7 | 3
score on a scale | 6.7 (6.7) | 8.7 (5.0)

6. Secondary Outcome: Mean Change From Baseline in Worst Stiffness Numeric Rating Scale (NRS) Score
Description: The Worst Stiffness NRS is a 1-item, self-administered questionnaire assessing the "worst" stiffness within the last 24 hours. The NRS for this item ranges from 0 (no stiffness) to 10 (stiffness as bad as you can imagine).
Time Frame: Week 12
Population: Worst Stiffness Numeric Rating Scale score was not assessed for 1 subject in the high dose group at week 12 as their assessments were not completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AMB-05X High Dose | AMB-05X Low Dose
Number analyzed (Participants) | 7 | 3
score on a scale | -2.4 (4.4) | -2.3 (1.5)

7. Secondary Outcome: Mean Change From Baseline in the Brief Pain Inventory (BPI) Pain Interference Index Score
Description: Brief Pain Inventory (BPI) Short Form is a self-administered questionnaire used to evaluate the severity of a subject's pain and the impact of this pain on the subject's daily functioning. The subject is asked to rate their worst, least, average, and current pain intensity, list current treatments and their perceived effectiveness, and rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a scale from 0 to 10, where higher scores mean more pain interference. The reported score is the mean of the seven interference items.
Time Frame: Week 12
Population: Brief Pain Inventory (BPI) Pain Interference Index Score was not assessed for 2 subjects in the high dose group at week 12 due to assessment not completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AMB-05X High Dose | AMB-05X Low Dose
Number analyzed (Participants) | 6 | 3
score on a scale | -2.8 (3.2) | -2.6 (1.8)

8. Secondary Outcome: EuroQol 5 Dimension 5 Level (EQ-5D-5L) Health Assessment
Description: EuroQol 5 Dimension 5 Level (EQ-5D-5L) is a widely used quality of life instrument that includes questions in each of 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate their health state by selecting the most appropriate statement in each of the five dimensions. Individual scores range from 1 to 5. The EQ-5D-5L scale score is the sum of the 5 individual EQ-5D-5L scores collected and ranges from 5 to 25. Lower scores represent a better quality of life.
Time Frame: Week 12
Population: EQ-5D-5L was not assessed for 1 subject in the high dose group at week 12 due to assessment not completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AMB-05X High Dose | AMB-05X Low Dose
Number analyzed (Participants) | 7 | 3
score on a scale | -0.9 (1.5) | -0.7 (1.5)

9. Secondary Outcome: Percentage of Subjects Who Respond With a Decrease of at Least 30% in Mean Brief Pain Inventory (BPI) Score
Description: The BPI Short Form is a self-administered questionnaire used to evaluate the severity of a subject's pain and the impact of this pain on the subject's daily functioning.
Time Frame: week 12
Population: Brief Pain Inventory Score was not assessed for 2 subjects in the high dose group at week 12 due to assessment not completed.
Measure: Count of Participants; unit: Participants
Groups:
- AMB-05X High Dose; AMB-05X Low Dose: Subjects received an intra-articular injection of AMB-05X once every 2 weeks for 12 weeks (for 6 treatments total).
Arm/Group | AMB-05X High Dose | AMB-05X Low Dose
Number analyzed (Participants) | 6 | 3
Participants | 5 | 2

10. Secondary Outcome: Serum Colony Stimulating Factor 1 (CSF1) Levels
Description: Serum CSF1 levels will be analyzed as a biomarker.
Time Frame: week 10
Population: Subjects with TGCT of the knee will receive intra-articular injection of AMB-05X once every 2 weeks for 12 weeks (for 6 treatments total). The results for serum CSF1 (pharmacodynamic data) concentrations were grouped by dose level (low or high Q2W) to better enable dose-response evaluation and treatment regimen optimization in continued clinical development.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- AMB-05X - Low Dose: Subjects with TGCT of the knee will receive intra-articular injection of a low dose of AMB-05X once every 2 weeks for 12 weeks (for 6 treatments total).
- AMB-05X - High Dose: Subjects with TGCT of the knee will receive intra-articular injection of high dose AMB-05X once every 2 weeks for 12 weeks (for 6 treatments total).
Arm/Group | AMB-05X - Low Dose | AMB-05X - High Dose
Number analyzed (Participants) | 3 | 8
pg/mL | 503 (725) | 1030 (301)

11. Secondary Outcome: Serum AMB-05X Levels
Description: Serum AMB-05X concentrations will be measured at Week 0 (pre-dose and 2 hours after the first dose), Week 2 (pre-dose [trough]), and Week 10 during steady state (including pre-dose [trough] and 2 hour after the last dose).
Time Frame: week 10
Population: Subjects with TGCT of the knee will receive intra-articular injection of AMB-05X once every 2 weeks for 12 weeks (for 6 treatments total). The results for serum AMB-05X (pharmacokinetic) concentrations were grouped by dose level (low or high Q2W) to better enable dose-response evaluation and treatment regimen optimization in continued clinical development.
Measure: Mean (Standard Deviation); unit: ug/ml
Groups:
- AMB-05X - Low Dose: Subjects with TGCT of the knee will receive intra-articular injection of low dose AMB-05X once every 2 weeks for 12 weeks (for 6 treatments total).
Arm/Group | AMB-05X - Low Dose | AMB-05X - High Dose
Number analyzed (Participants) | 3 | 8
ug/ml | 2.1 (3.2) | 33.0 (31.5)

12. Secondary Outcome: Serum Anti-AMB-05X Antibody Levels
Description: Anti-drug antibody (ADA) analysis will also be performed on select serum samples.
Time Frame: week 10
Population: Subjects with TGCT of the knee will receive intra-articular injection of AMB-05X once every 2 weeks for 12 weeks (for 6 treatments total). The results for serum anti-drug antibody development were grouped by dose level (low or high Q2W) to better enable dose-response evaluation and treatment regimen optimization in continued clinical development.
Measure: Count of Participants; unit: Participants
Arm/Group | AMB-05X - Low Dose | AMB-05X - High Dose
Number analyzed (Participants) | 3 | 8
Participants
  Pts ADA positive at any visit analyzed | 0 | 0
  Pts ADA negative at all visits analyzed | 3 | 8

13. Secondary Outcome: Synovial Fluid CSF1
Description: Measurement of CSF1 in synovial fluid (pharmacodynamic marker)
Time Frame: Week 10
Population: Subjects with TGCT of the knee will receive intra-articular injection of AMB-05X once every 2 weeks for 12 weeks (for 6 treatments total). The results for synovial CSF1 (pharmacodynamic data) concentrations were grouped by dose level (low or high Q2W) to better enable dose-response evaluation and treatment regimen optimization in continued clinical development. In the low-dose arm, 1 subject had sufficient samples to analyze.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | AMB-05X - Low Dose | AMB-05X - High Dose
Number analyzed (Participants) | 1 | 8
ng/ml | 37.1 (NA) — As data are reported for 1 subject only, no SD can be calculated. | 22.6 (3.1)

14. Secondary Outcome: Synovial AMB-05X Levels
Description: Synovial AMB-05X concentrations will be measured at Weeks 0, 2, 4, 6, 8, and 10 (all at pre-dose [trough]).
Time Frame: Week 10
Population: Subjects with TGCT of the knee will receive intra-articular injection of AMB-05X once every 2 weeks for 12 weeks (for 6 treatments total). Results for synovial AMB-05X (pharmacokinetic data) were grouped by dose level (low or high Q2W) to better enable dose-response evaluation and treatment regimen optimization in continued clinical development. In the low-dose arm, 1 subject had sufficient samples for analysis.
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | AMB-05X - Low Dose | AMB-05X - High Dose
Number analyzed (Participants) | 1 | 8
ug/ml | 36.3 (NA) — As data are reported for 1 subject only, no SD can be calculated. | 153 (138)

15. Secondary Outcome: Synovial Anti-AMB-05X Antibody (ADA) Levels
Description: Anti-drug antibody (ADA) analysis will also be performed on select synovial samples.
Time Frame: Week 10
Population: Subjects with TGCT of the knee who receive intra-articular injection of AMB-05X once every 2 weeks for 12 weeks (for 6 treatments total). Results for synovial anti-drug antibody development are grouped by dose level (low or high Q2W) to better enable dose-response evaluation and treatment regimen optimization in continued clinical development.
Measure: Number; unit: participants
Arm/Group | AMB-05X - Low Dose | AMB-05X - High Dose
Number analyzed (Participants) | 3 | 8
participants
  Pts ADA positive at any visit analyzed | 1 | 0
  Pts ADA negative at all visits analyzed | 2 | 8

16. Secondary Outcome: Proportions of Subjects Who Achieved Objective Response as Their Best Overall Tumor Response, Per Modified Response Evaluation Criteria in Solid Tumors (RECIST).
Description: Objective response was measured using the modified Response Evaluation Criteria in Solid Tumors (RECIST), which requires >/=30% reduction in the sum of short-axis diameters of 2 target lesions.
Time Frame: 12 Weeks
Population: All enrolled patients
Measure: Count of Participants; unit: Participants
Arm/Group | AMB-05X High Dose | AMB-05X Low Dose
Number analyzed (Participants) | 8 | 3
Participants | 4 | 1

ADVERSE EVENTS:
Time Frame: up to 24 weeks
Groups:
- AMB-05X High Dose; AMB-05X Low Dose: Subjects received an injection of AMB-05X once every 2 weeks for 12 weeks (for 6 treatments total).
Arm/Group | AMB-05X High Dose | AMB-05X Low Dose
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/3
Other Adverse Events (participants affected / at risk) | 7/8 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AMB-05X High Dose (N=8) | AMB-05X Low Dose (N=3)
Fatigue (General disorders) | 4 | 1
Face Edema (General disorders) | 4 | 0
peripheral edema (General disorders) | 3 | 0
localised edema (General disorders) | 2 | 0
periorbital edema (Eye disorders) | 5 | 0
arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
rash (Skin and subcutaneous tissue disorders) | 4 | 0
pruritis (Skin and subcutaneous tissue disorders) | 2 | 1
paresthesia (Nervous system disorders) | 2 | 0
COVID-19 (Infections and infestations) | 2 | 1
hypertension (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT04731675/Prot_SAP_000.pdf